CLINICAL TRIAL: NCT00726453
Title: A Clinical Evaluation of the Medtronic Resolute Zotarolimus-Eluting Coronary Stent System in the Treatment of De Novo Lesions in Native Coronary Arteries With a Reference Vessel Diameter of 2.25 mm to 4.2mm
Brief Title: The Medtronic RESOLUTE US Clinical Trial
Acronym: R-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP102
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Artery Disease
Keywords: TARGET VESSEL REVASCULARIZATION (TVR); MYOCARDIAL INFARCTION (MI); TARGET VESSEL FAILURE (TVF); TARGET LESION REVASCULARIZATION (TLR); TARGET LESION FAILURE (TLF); STENT THROMBOSIS; RESTENOTIC LESION; PERCUTANEOUS CORONARY INTERVENTION (PCI)
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resolute Zotarolimus-Eluting Coronary Stent (Experimental): Implantation of a Resolute Zotarolimus-Eluting Coronary Stent
  Interventions: Device: Resolute Zotarolimus-Eluting Coronary Stent

INTERVENTIONS:
Device: Resolute Zotarolimus-Eluting Coronary Stent — Implantation of a Resolute Zotarolimus-Eluting Coronary Stent

SUMMARY:
The objective of the study is to assess the safety and effectiveness of the Resolute Zotarolimus-Eluting Coronary Stent System for the treatment of de novo lesions in native coronary arteries with a reference vessel diameter (RVD) of 2.25 mm to 4.2 mm.

DETAILED DESCRIPTION:
The trial is comprised of four studies: the 2.25 mm - 3.5 mm main study (1242 patients), the 2.25 mm - 3.5 mm Angio/IVUS sub-study (100 patients), the 4.0 mm sub-study (60 patients), and the 38 mm Length Sub-study (114 patients). A patient's inclusion in a given study is dependent on the size (diameter or length) of the stent(s) the patient receives.

ELIGIBILITY:
General and Angiographic Inclusion Criteria highlights:

* Acceptable candidate for percutaneous coronary intervention (PCI),stenting, and emergency coronary artery bypass graft surgery
* Clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia and/or positive functional study
* Informed consent
* Patient agrees to comply with specified follow-up evaluations at same investigational site
* Single target lesion or two target lesions located in separate coronary arteries
* De novo lesion(s) in native coronary artery(ies)
* Target lesion(s) ≤ 27 mm in length (or ≤ 35 mm for a lesion to be treated with a 38 mm length stent)
* Target vessel(s) have reference vessel diameter 2.25 mm to 4.2 mm, (or 3.0 to 4.2 mm for it to be treated with a 38 mm length stent)

General and Angiographic Exclusion Criteria highlights:

* Within 7 days of implant platelet count <100,000 cells/mm³ or >700,000 cells/mm³; WBC count <3,000 cells/mm³; serum creatinine level >2.5 mg/dl
* Acute MI within 72 hrs of the index procedure (QWMI or any elevation of CK-MB > lab upper limit of normal)
* Previous PCI of target vessel(s) within 9 months prior to the procedure
* Planned PCI of any vessel within 30 days post-index procedure and/or planned PCI of target vessel(s) within 12 months post-index procedure
* History of stroke or TIA within prior 6 months
* Participating in investigational drug/device study that has not completed primary endpoint or interferes with study endpoints
* Inability to comply with required trial antiplatelet regimen
* Previous stent in target vessel unless it has been at least 9 months since stent placed and target lesion(s) is/are at least 15 mm from previous stent
* Target vessel(s) has/have other lesions w/ > 40% diameter stenosis
* Unprotected left main coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1516 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Principal Investigator — Columbia University College of Physicians & Surgeons; Laura Mauri, MD, MSc, Principal Investigator — Brigham and Women's Hospital; Alex C Yeung, MD, Principal Investigator — Stanford University
Locations (1):
- East Texas Medical Center, Tyler, Texas, United States

REFERENCES:
- [Derived] Silber S, Kirtane AJ, Belardi JA, Liu M, Brar S, Rothman M, Windecker S. Lack of association between dual antiplatelet therapy use and stent thrombosis between 1 and 12 months following resolute zotarolimus-eluting stent implantation. Eur Heart J. 2014 Aug 1;35(29):1949-56. doi: 10.1093/eurheartj/ehu026. Epub 2014 Feb 7. PMID 24510638
- [Derived] Silber S, Serruys PW, Leon MB, Meredith IT, Windecker S, Neumann FJ, Belardi J, Widimsky P, Massaro J, Novack V, Yeung AC, Saito S, Mauri L. Clinical outcome of patients with and without diabetes mellitus after percutaneous coronary intervention with the resolute zotarolimus-eluting stent: 2-year results from the prospectively pooled analysis of the international global RESOLUTE program. JACC Cardiovasc Interv. 2013 Apr;6(4):357-68. doi: 10.1016/j.jcin.2012.11.006. Epub 2013 Mar 20. PMID 23523454
- [Derived] Farooq V, Vranckx P, Mauri L, Cutlip DE, Belardi J, Silber S, Widimsky P, Leon M, Windecker S, Meredith I, Negoita M, van Leeuwen F, Neumann FJ, Yeung AC, Garcia-Garcia HM, Serruys PW. Impact of overlapping newer generation drug-eluting stents on clinical and angiographic outcomes: pooled analysis of five trials from the international Global RESOLUTE Program. Heart. 2013 May;99(9):626-33. doi: 10.1136/heartjnl-2012-303368. Epub 2013 Mar 6. PMID 23468513
- [Derived] Mauri L, Leon MB, Yeung AC, Negoita M, Keyes MJ, Massaro JM. Rationale and design of the clinical evaluation of the Resolute Zotarolimus-Eluting Coronary Stent System in the treatment of de novo lesions in native coronary arteries (the RESOLUTE US clinical trial). Am Heart J. 2011 May;161(5):807-14. doi: 10.1016/j.ahj.2011.03.015. Epub 2011 Mar 29. PMID 21570508
- [Derived] Yeung AC, Leon MB, Jain A, Tolleson TR, Spriggs DJ, Mc Laurin BT, Popma JJ, Fitzgerald PJ, Cutlip DE, Massaro JM, Mauri L; RESOLUTE US Investigators. Clinical evaluation of the Resolute zotarolimus-eluting coronary stent system in the treatment of de novo lesions in native coronary arteries: the RESOLUTE US clinical trial. J Am Coll Cardiol. 2011 Apr 26;57(17):1778-83. doi: 10.1016/j.jacc.2011.03.005. Epub 2011 Apr 4. PMID 21470813
- See also: Medtronic Home Page — http://www.medtronic.com
- See also: Medtronic Clinical Trials Link — http://clinicaltrials.medtronic.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Enrollment Group: All patients may have one or two lesions, if the two lesions are located in separate coronary arteries. Patients were assigned in to one of four sub-studies based on the stent required:
  2.25 mm - 3.5 mm Main study, 2.25 mm - 3.5 mm Angio/IVUS Sub-study, 4.0 mm Sub-study, or 38 mm Length Sub-study.
  Patients enrolled in the 2.25 - 3.5 mm Main Study, the 2.25 mm - 3.5 mm Angio/IVUS Sub-study, and the 4.0 mm Sub-study are collectively referred to as the Primary Enrollment Group (PEG).
- 38 mm Length Sub-study: All patients may have one or two lesions, if the two lesions are located in separate coronary arteries. Patients were assigned in to one of four sub-studies based on the stent required this group is the 38 mm Length Main study. Enrollment in this group opened after the Primary Enrollment Group had closed.
Period: Primary Enrollment Group
Arm/Group | Primary Enrollment Group | 38 mm Length Sub-study
Started | 1402 | 0
Completed | 1371 | 0
Not Completed | 31 | 0
Not completed — Death | 18 | 0
Not completed — Withdrawal by Subject | 13 | 0
Period: 38 mm Length Group
Arm/Group | Primary Enrollment Group | 38 mm Length Sub-study
Started | 0 | 114
Completed | 0 | 111 (This sub-study completed the primary endpoint in March 2012 results not yet available.)
Not Completed | 0 | 3
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- 38 mm Length Sub-study: All patients may have one or two lesions, if the two lesions are located in separate coronary arteries. Patients were assigned in to one of four sub-studies based on the stent required this group is the 38 mm Length Main study. Enrollment in this group opened after the Primary Enrollment Group had closed. This sub-study completed the primary endpoint in March 2012 results not yet available.
- Total: Total of all reporting groups
Arm/Group | Primary Enrollment Group | 38 mm Length Sub-study | Total
Number analyzed (Participants) | 1402 | 114 | 1516
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (10.7) | 64.8 (9.7) | 64.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 444 | 30 | 474
  Male | 958 | 84 | 1042
Region of Enrollment [Number; unit: participants]
  United States | 1402 | 114 | 1516

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure (TLF)
Description: Target Lesion Failure (TLF) at 12 months post-procedure, defined as Cardiac Death, Target Vessel Myocardial Infarction (TVMI) (Q wave and non-Q wave) or clinically-driven Target Lesion Revascularization (TLR) by percutaneous or surgical methods.
Time Frame: 12 Months
Measure: Number; unit: percentage of participants
Arm/Group | Primary Enrollment Group
Number analyzed (Participants) | 1376
percentage of participants | 4.7

2. Secondary Outcome: Target Vessel Failure (TVF)
Description: Target Vessel Failure (TVF) composite endpoint and each individual component (Cardiac Death, Target Vessel MI, or clinically-driven Target Vessel Revascularization (TVR) by percutaneous or surgical methods).
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Primary Enrollment Group
Number analyzed (Participants) | 1376
percentage of participants | 6.3

3. Secondary Outcome: Major Adverse Cardiac Event (MACE)
Description: Major Adverse Cardiac Event (MACE) composite endpoint and each individual component (death, Target Vessel MI (Q wave and non-Q wave), emergent coronary bypass surgery (CABG), or clinically-driven repeat Target Lesion Revascularization (TLR) by percutaneous or surgical methods).
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Primary Enrollment Group
Number analyzed (Participants) | 1376
percentage of participants | 5.5

4. Secondary Outcome: Death
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Primary Enrollment Group
Number analyzed (Participants) | 1376
percentage of participants | 1.3

5. Secondary Outcome: Target Vessel MI
Description: Target Vessel MI (as determined by extended historical and ARC definitions).
Time Frame: 12 months
Measure: Number; unit: percentage of eligible participants
Arm/Group | Primary Enrollment Group
Number analyzed (Participants) | 1376
percentage of eligible participants | 1.4

6. Secondary Outcome: Stent Thrombosis (ST)
Description: Stent Thrombosis (ST) (as determined by historic and ARC definitions).
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Primary Enrollment Group
Number analyzed (Participants) | 1376
percentage of participants | 0.1

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Primary Enrollment Group: All patients may have one or two lesions, if the two lesions are located in separate coronary arteries. Patients were assigned in to one of four sub-studies based on the stent required:
  2.25 mm - 3.5 mm Main study, 2.25 mm - 3.5 mm Angio/IVUS Sub-study, 4.0 mm Sub-study and are collectively referred to as the Primary Enrollment Group (PEG).
Arm/Group | Primary Enrollment Group | 38 mm Length Sub-Study
Serious Adverse Events (participants affected / at risk) | 509/1402 | 71/114
Other Adverse Events (participants affected / at risk) | 724/1402 | 67/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Enrollment Group (N=1402) | 38 mm Length Sub-Study (N=114)
Anaemia (Blood and lymphatic system disorders) | 12 (16) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 3 (3) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 21 (21) | 3 (3)
Angina Pectoris (Cardiac disorders) | 68 (83) | 6 (6)
Angina Unstable (Cardiac disorders) | 19 (19) | 2 (2)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm Coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 17 (20) | 2 (3)
Atrial Flutter (Cardiac disorders) | 3 (3) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 18 (21) | 3 (7)
Cardiac Valve Disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 56 (60) | 11 (12)
Coronary Artery Dissection (Cardiac disorders) | 13 (13) | 7 (7)
Coronary Artery Embolism (Cardiac disorders) | 0 (0) | 2 (2)
Coronary Artery Occlusion (Cardiac disorders) | 2 (2) | 1 (1)
Coronary Artery Perforation (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Restenosis (Cardiac disorders) | 12 (12) | 2 (2)
Coronary Artery Stenosis (Cardiac disorders) | 13 (14) | 1 (1)
In-Stent Coronary Artery Restenosis (Cardiac disorders) | 13 (14) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 7 (7) | 2 (2)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 3 (3) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 4 (5) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 4 (4) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hyperparathyroidism Primary (Endocrine disorders) | 1 (1) | 0 (0)
Amaurosis Fugax (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 3 (5)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eye Swelling (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 10 (13) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's Oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 21 (23) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 3 (4) | 1 (1)
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 2 (5) | 0 (0)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 3 (4) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Splenic Artery Aneurysm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Adverse Drug Reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Catheter Site Haemorrhage (General disorders) | 2 (2) | 0 (0)
Chest Discomfort (General disorders) | 7 (8) | 0 (0)
Chest Pain (General disorders) | 79 (98) | 7 (7)
Death (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Granuloma (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Implant Site Effusion (General disorders) | 1 (1) | 0 (0)
Injection Site Haematoma (General disorders) | 2 (2) | 1 (1)
Injection Site Haemorrhage (General disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 2 (2) | 0 (0)
Multi-Organ Failure (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 32 (39) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder Disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0)
Abscess Neck (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Catheter Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Cellulitis Staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Clostridial Infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 5 (8) | 0 (0)
Endocarditis Bacterial (Infections and infestations) | 1 (2) | 0 (0)
Escherichia Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 9 (13) | 0 (0)
Liver Abscess (Infections and infestations) | 1 (1) | 0 (0)
Perirectal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 20 (20) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic Shock (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Syphilitic Endocarditis Of Heart Valve (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous Graft Thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Lesion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Stent Occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombosis In Device (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urethral Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Mb Increased (Investigations) | 2 (2) | 0 (0)
Blood Creatinine Increased (Investigations) | 2 (2) | 0 (0)
Blood Glucose Increased (Investigations) | 1 (1) | 0 (0)
Cardiac Enzymes Increased (Investigations) | 7 (7) | 3 (3)
Cardiac Stress Test Abnormal (Investigations) | 2 (2) | 0 (0)
Ejection Fraction Decreased (Investigations) | 1 (1) | 0 (0)
Troponin T Increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone Lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 (12) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Bronchioloalveolar Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Choroid Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 13 (14) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 14 (14) | 1 (1)
Cervical Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Nerve Compression (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 4 (4) | 0 (0)
Syncope (Nervous system disorders) | 9 (10) | 3 (3)
Syncope Vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 5 (6) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 2 (2) | 1 (1)
Bladder Neck Sclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (7) | 0 (0)
Haemorrhage Urinary Tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 0 (0)
Nephrotic Syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal Failure (Renal and urinary disorders) | 11 (11) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hypoaesthesia Facial (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Carotid Endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary Revascularisation (Surgical and medical procedures) | 6 (7) | 1 (1)
Hip Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Hysterosalpingo-Oophorectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical Device Implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal Artery Stent Placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Therapeutic Embolisation (Surgical and medical procedures) | 1 (1) | 1 (1)
Accelerated Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 3 (3) | 0 (0)
Arterial Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial Stenosis Limb (Vascular disorders) | 1 (2) | 0 (0)
Arteriovenous Fistula (Vascular disorders) | 0 (0) | 1 (1)
Artery Dissection (Vascular disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 2 (3) | 0 (0)
Femoral Arterial Stenosis (Vascular disorders) | 3 (5) | 0 (0)
Femoral Artery Occlusion (Vascular disorders) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 13 (14) | 1 (1)
Hypotension (Vascular disorders) | 12 (12) | 0 (0)
Iliac Artery Stenosis (Vascular disorders) | 2 (2) | 0 (0)
Intermittent Claudication (Vascular disorders) | 6 (7) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 3 (7) | 1 (1)
Peripheral Vascular Disorder (Vascular disorders) | 7 (8) | 2 (2)
Poor Peripheral Circulation (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Subclavian Steal Syndrome (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular Pseudoaneurysm (Vascular disorders) | 3 (4) | 0 (0)
Venous Insufficiency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Enrollment Group (N=1402) | 38 mm Length Sub-Study (N=114)
Angina Pectoris (Cardiac disorders) | 171 (212) | 16 (20)
Nausea (Gastrointestinal disorders) | 0 (0) | 10 (10)
Chest Pain (General disorders) | 204 (256) | 23 (32)
Fatigue (General disorders) | 0 (0) | 8 (8)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 10 (11)
Oedema (General disorders) | 0 (0) | 6 (6)
Oedema Peripheral (General disorders) | 0 (0) | 9 (11)
Back Pain (Musculoskeletal and connective tissue disorders) | 92 (99) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 77 (81) | 17 (18)
Dizziness (Nervous system disorders) | 74 (79) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 106 (113) | 13 (15)
Hypertension (Vascular disorders) | 0 (0) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other